CLINICAL TRIAL: NCT06165497
Title: Short Practices Well-being Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-1324; Protocol Version 11/20/2023 (Other: UW- Madison); A171600 (Other: UW- Madison); EDUC/COUNSELING PSYCH (Other: UW- Madison)
Record Dates: First submitted 2023-11-28; First posted 2023-12-11 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Well-Being, Psychological
Keywords: meditation; mobile health; mindfulness; self-compassion; gratitude
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Mindfulness, 5 minutes, male voice (Experimental): Mindfulness meditation, 5 minutes duration, with a male speaker.
  Interventions: Behavioral: Meditation practices
- Mindfulness, 10 minutes, male voice (Experimental): Mindfulness meditation, 10 minutes duration, with a male speaker.
  Interventions: Behavioral: Meditation practices
- Mindfulness, 5 minutes, female voice (Experimental): Mindfulness meditation, 5 minutes duration, with a female speaker.
  Interventions: Behavioral: Meditation practices
- Mindfulness, 10 minutes, female voice (Experimental): Mindfulness meditation, 10 minutes duration, with a female speaker.
  Interventions: Behavioral: Meditation practices
- Self-compassion, 5 minutes, male voice (Experimental): Self-compassion meditation, 5 minutes duration, with a male speaker.
  Interventions: Behavioral: Meditation practices
- Self-compassion, 10 minutes, male voice (Experimental): Self-compassion meditation, 10 minutes duration, with a male speaker.
  Interventions: Behavioral: Meditation practices
- Self-compassion, 5 minutes, female voice (Experimental): Self-compassion meditation, 5 minutes duration, with a female speaker.
  Interventions: Behavioral: Meditation practices
- Self-compassion, 10 minutes, female voice (Experimental): Self-compassion meditation, 10 minutes duration, with a female speaker.
  Interventions: Behavioral: Meditation practices
- Gratitude, 5 minutes, male voice (Experimental): Gratitude meditation, 5 minutes duration, with a male speaker.
  Interventions: Behavioral: Meditation practices
- Gratitude, 10 minutes, male voice (Experimental): Gratitude meditation, 10 minutes duration, with a male speaker.
  Interventions: Behavioral: Meditation practices
- Gratitude, 5 minutes, female voice (Experimental): Gratitude meditation, 5 minutes duration, with a female speaker.
  Interventions: Behavioral: Meditation practices
- Gratitude, 10 minutes, female voice (Experimental): Gratitude meditation, 10 minutes duration, with a female speaker.
  Interventions: Behavioral: Meditation practices
- Internet-as-usual, 5 minutes (Other): Participants will be instructed to use the internet as they typical do for 5 minutes.
  Interventions: Other: Internet-as-usual
- Internet-as-usual, 10 minutes (Other): Participants will be instructed to use the internet as they typical do for 10 minutes.
  Interventions: Other: Internet-as-usual

INTERVENTIONS:
Behavioral: Meditation practices — Participants will listen to recordings of short meditation practices drawn from the Healthy Minds Program.
  Arms: Gratitude, 10 minutes, female voice; Gratitude, 10 minutes, male voice; Gratitude, 5 minutes, female voice; Gratitude, 5 minutes, male voice; Mindfulness, 10 minutes, female voice; Mindfulness, 10 minutes, male voice; Mindfulness, 5 minutes, female voice; Mindfulness, 5 minutes, male voice; Self-compassion, 10 minutes, female voice; Self-compassion, 10 minutes, male voice; Self-compassion, 5 minutes, female voice; Self-compassion, 5 minutes, male voice
Other: Internet-as-usual — Participants will be instructed to use the internet as they typically do.
  Arms: Internet-as-usual, 10 minutes; Internet-as-usual, 5 minutes

SUMMARY:
The goal of this research study is to better understand the effects of short practices on well-being.

Participants will be asked to complete a task that will take 5-10 minutes, followed by a set of surveys. They will also be invited to complete a second set of surveys ~7 days later.

DETAILED DESCRIPTION:
The aim of this study is to better understand the effects of short practices on well-being. In the initial part of the study, participants will be required to complete a set of surveys assessing their health along with demographic measures. Participants will also be asked to complete a brief task. They will be asked sensitive questions (e.g., about your psychological state, mental health). To have their submission accepted, participants must correctly answer questions designed to check if they are paying attention. This part of the study will take approximately 24 minutes to complete. Anonymized data may be made available to other researchers. One week after completing this study, participants will be invited to complete a second set of surveys.

ELIGIBILITY:
Inclusion Criteria:

* United States and United Kingdom residents 18 year or older

Exclusion Criteria:

* Inability or unwillingness to complete the study
* Fail to pass the attention check embedded in the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5049 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Affect Schedule Positive Affect | Current positive affect pre- and post- short tasks (up to 10 minutes).
  Participants respond to a 10-item survey indicating their current mood. Response options range from 1 (very slightly or not at all) to 5 (extremely). Five items reflect positive affect. Higher scores indicate higher positive affect.
Positive and Negative Affect Schedule Negative Affect | Current negative affect pre- and post- short tasks (up to 10 minutes).
  Participants respond to a 10-item survey indicating their current mood. Response options range from 1 (very slightly or not at all) to 5 (extremely). Five items reflect negative affect. Higher scores indicate higher negative affect.

SECONDARY OUTCOMES:
State Mindfulness Scale | Up to 10 minutes
  Participants respond to a 21-item survey indicating their state mindfulness. Response options range from 1 (not at all) to 5 (very well). Higher scores indicate higher state mindfulness.
State Self-Compassion Scale Short Form | Up to 10 minutes
  Participants respond to a 6-item survey indicating their state self-compassion. Response options range from 1 (not at all true for me) to 5 (very true for me). Higher scores indicate higher state self-compassion.
Gratitude Adjective Checklist - 3 | Up to 10 minutes
  Participants respond to a 3-item survey indicating their state gratitude. Response options range from 1 (not at all) to 5 (extremely). Higher scores indicate higher state gratitude.
Adverse reaction to short tasks | Up to 10 minutes
  Participants will indicate whether they had a "distressing experience" (yes/no) during the task they completed.
Meditation practice using the short task practice type. | 7-day follow-up
  Participants will be asked how many days they practiced the three meditation practice types during the past week.
Healthy Minds Program download | 7-day follow-up
  Participants will be asked whether they downloaded the Healthy Minds Program and how many days they used the app if they downloaded it.
Ruminative Response Style | Pre- short tasks and 7-day follow-up
  Participants respond to an 8-item survey indicating their level of rumination. Response options range from 1 (almost never) to 4 (almost always). Higher scores indicate higher rumination.
NIH Toolbox Loneliness | Pre- short tasks and 7-day follow-up
  Participants respond to a 5-item survey indicating their level of loneliness. Response options range from 1 (never) to 5 (always). Higher scores indicate higher loneliness.
Perceived Stress Scale | Pre- short tasks and 7-day follow-up
  Participants respond to a 4-item survey indicating their level of perceived stress. Response options range from 1 (never) to 5 (very often). Higher scores indicate higher perceived stress.
PROMIS Anxiety | Pre- short tasks and 7-day follow-up
  Participants respond to a 4-item survey indicating their level of anxiety. Response options range from 1 (never) to 5 (always). Higher scores indicate higher anxiety.
PROMIS Depression | Pre- short tasks and 7-day follow-up
  Participants respond to a 4-item survey indicating their level of depression. Response options range from 1 (never) to 5 (always). Higher scores indicate higher depression.
Self-Compassion Scale Short Form | Pre- short tasks and 7-day follow-up
  Participants respond to a 12-item survey indicating their level of trait self-compassion. Response options range from 1 (almost never) to 5 (almost always). Higher scores indicate higher trait self-compassion.
Five Facet Mindfulness Questionnaire Short Form | Pre- short tasks and 7-day follow-up
  Participants respond to a 15-item survey indicating their level of trait mindfulness. Response options range from 1 (never or very rarely true) to 5 (very often or always true). Higher scores indicate higher trait mindfulness.
Gratitude Questionnaire | Pre- short tasks and 7-day follow-up
  Participants respond to a 6-item survey indicating their level of trait gratitude. Response options range from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate higher trait gratitude.
Positive and Negative Affect Schedule Positive Affect | 7-day follow-up
  Participants respond to a 10-item survey indicating their current mood. Response options range from 1 (very slightly or not at all) to 5 (extremely). Five items reflect positive affect. Higher scores indicate higher positive affect.
Positive and Negative Affect Schedule Negative Affect | 7-day follow-up
  Participants respond to a 10-item survey indicating their current mood. Response options range from 1 (very slightly or not at all) to 5 (extremely). Five items reflect negative affect. Higher scores indicate higher negative affect.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Goldberg, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No